CLINICAL TRIAL: NCT01476904
Title: A 3-month Safety Evaluation Extension to the 12-week E004-C Study in Asthma Patients (A Double Blinded, Placebo-controlled, Parallel, 3-month Safety Study in Adolescent and Adult Patients With Asthma)
Brief Title: Safety Study in Adolescent and Adult Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: API-E004-CL-C2
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Asthma; Shortness of breath
MeSH Terms: conditions — Asthma; Dyspnea | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm T (Experimental): Arm T is the experimental treatment arm consisting of 2 x 125 mcg/inhalations of epinephrine inhalation, QID, with 4-6 hr intervals
  Interventions: Drug: Epinephrine inhalation
- Arm P (Placebo Comparator): Arm P is a placebo comparator consisting of 2× 0 mcg of placebo inhalations, QID, with 4-6 hr intervals
  Interventions: Drug: Placebo
- Arm A (Active Comparator): Arm A is an active comparator, Primatene Mist, consisting of 2× 220 mcg/inhalation, QID, with 4-6 hr intervals
  Interventions: Drug: Primatene Mist

INTERVENTIONS:
Drug: Placebo — 0 mcg/inhalation, 2 inhalations QID
  Arms: Arm P
Drug: Primatene Mist — 220 mcg/inhalation, 2 inhalations QID
  Arms: Arm A
Drug: Epinephrine inhalation — 125 mcg/inhalation, 2 inhalations QID
  Arms: Arm T

SUMMARY:
E004-C2 is a continuation of E004-C for safety evaluations with additional 3 months to be able to assess the 6-month safety profile for E004 (epinephrine inhalation) versus placebo in a double-blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who have successfully completed the E004-C study within the last 135 days or those who are actively enrolled in the current study E004-C at the time of the study extension initiation
* Male and female asthma patients aged 12 - 75 years
* Patients with documented asthma, requiring inhaled epinephrine or beta 2-agonist treatment
* No significant changes in asthma therapy and no asthma-related hospitalization or emergency visits, within 4 weeks prior to Screening
* Demonstrating satisfactory techniques in the use of metered-dose inhaler and a hand held peak expiratory flow meter
* Female patients of child-bearing potential must be non-pregnant and non-lactating at Screening and throughout the study, and must use an acceptable method of contraception during the study

Exclusion Criteria:

* A smoking history of 10-pack years, or having smoked within 12 months of screening
* Any current or past medical conditions that, per investigator discretion, might significantly affect responses to the study drugs, other than asthma
* Concurrent clinically significant diseases
* Known intolerance or hypersensitivity to any component of the study drugs
* Recent infection of the respiratory tract, before screening
* Use of prohibited medications
* Having been on other investigational drug/device studies in the last 30 days prior to screening
* Known or highly suspected substance abuse

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events | up to 12 weeks
  Recording of all adverse events experienced during the course of the study

SECONDARY OUTCOMES:
Change in 12 lead ECG including QT/QTc analysis | Study visit 4, 8 and 12, greater than one hour after last dose
  A 12-lead ECG (routine and QT/QTc) will be measured and recorded, provided that dosing of study drug has been performed greater than 1 hour prior to conducting the measurements.
Asthma Exacerbations | up to 12 weeks
  Review use of resuce inhaler for treatment of asthma exacrbations occuring between doses of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Safety Monitor, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (27):
- United States (27):
  - Amphastar Site 0006, Costa Mesa, California
  - Amphastar Site 0005, Los Angeles, California
  - Amphastar Site 0004, Orange, California
  - Amphastar Site 0001, San Jose, California
  - Amphastar Site 0003, Stockton, California
  - Amphastar Site 0008, Denver, Colorado
  - Amphastar Site 0009, Wheat Ridge, Colorado
  - Amphastar Site 0011, Iowa City, Iowa
  - Amphastar Site 0013, North Dartmouth, Massachusetts
  - Amphastar Site 0014, Minneapolis, Minnesota
  - Amphastar Site 0015, Plymouth, Minnesota
  - Amphastar Site 0016, St Louis, Missouri
  - Amphastar Site 0017, Bozeman, Montana
  - Amphastar Site 0019, Bellevue, Nebraska
  - Amphastar Site 0020, Skillman, New Jersey
  - Amphastar Site 0018, Raleigh, North Carolina
  - Amphastar Site 0021, Cincinnati, Ohio
  - Amphastar Site 0024, Ashland, Oregon
  - Amphastar Site 0022, Eugene, Oregon
  - Amphastar Site 0023, Lake Oswego, Oregon
  - Amphastar Site 0025, Medford, Oregon
  - Amphastar Site 0026, Portland, Oregon
  - Amphastar Site 0029, North Charleston, South Carolina
  - Amphastar Site 0031, El Paso, Texas
  - Amphastar Site 0030, New Braunfels, Texas
  - Amphastar Site 0033, Richmond, Virginia
  - Amphastar Site 0034, Seattle, Washington

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Derived] Kerwin EM, Tashkin DP, Korenblat PE, Greos LS, Pearlman DS, Bensch GW, Miller SD, Marrs T, Luo MZ, Zhang JY. Long-term safety and efficacy studies of epinephrine HFA metered-dose inhaler (Primatene(R) Mist): a two-stage randomized controlled trial. J Asthma. 2021 May;58(5):633-644. doi: 10.1080/02770903.2020.1713147. Epub 2020 Jan 20. PMID 31959019